CLINICAL TRIAL: NCT01791088
Title: A Pharmacodynamic Study of Sirolimus in Older Children and Adults With Advanced Solid Malignancies
Brief Title: Sirolimus in Treating Patients With Solid Tumors That Are Metastatic or Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1169; NCI-2012-01166 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (sirolimus) (Experimental): Patients receive sirolimus PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sirolimus; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sirolimus — Given PO
  Other Names: AY 22989; Rapamune; rapamycin; SLM
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies sirolimus in treating patients with solid tumors that are metastatic or cannot be removed by surgery. Sirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the magnitude, inter-individual variability and time course of sirolimus-induced changes in fasting serum glucose and triglycerides.

SECONDARY OBJECTIVES:

I. To assess candidate genetic variants for their correlation with changes in fasting glucose and/or triglycerides.

II. To assess tumor response by the Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) and explore whether there is any correlation between response and changes in fasting glucose and/or triglycerides.

III. To assess toxicity by the Common Terminology Criteria for Adverse Events (CTCAE, version 4.0) and explore whether there is any correlation between toxicities and changes in fasting glucose and/or triglycerides.

IV. To quantify and determine the functional status of circulating regulatory T cells (Tregs) before and during treatment.

OUTLINE:

Patients receive sirolimus orally (PO) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Weight >= 40 kg
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy > 3 months
* Absolute neutrophil count (ANC) >= l500/ul
* Hemoglobin >= 9g/dL
* Platelets >= 100,000/ ul
* Total bilirubin < 1.5 x upper limit of normal
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvate transaminase (SGPT) < 2.5 x upper limit of normal for patients without liver metastases OR SGOT and SGPT < 5 x upper limit of normal for patients with liver metastases
* Measurable or non-measurable disease will be allowed
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, up until 30 days after final study treatment; should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients taking substrates, inhibitors, or inducers of cytochrome P450 (CYP)3A4 should be encouraged to switch to alternative drugs whenever possible, given the potential for drug-drug interactions with sirolimus
* Signed informed consent

Exclusion Criteria:

* Prior treatment with a mammalian target of rapamycin (mTOR) inhibitor (including sirolimus) is allowed; however, patients with >= grade 3 toxicities with an mTOR inhibitor are excluded
* Fasting glucose > 126 mg/dL or fasting triglycerides > 150 mg/dL; patients are allowed to be on oral anti-hyperglycemic and anti-lipid therapies, but cannot be on insulin
* Patients who have had chemotherapy or immunotherapy within 3 weeks of starting study drug, or radiotherapy within 14 days of starting study drug, or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents or any concomitant antineoplastic therapy, with the exception of androgen ablating agents (for patients with prior prostate cancer)
* Serious underlying medical or psychiatric illnesses that would, in the opinion of the treating physician, substantially increase the risk for complications related to treatment; similarly, any unstable medical condition that in the opinion of the treating physician or study investigators, would interfere with determination of the study objectives
* Pregnancy or breastfeeding
* Major surgery within 4 weeks

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-06-13 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Change in fasting glucose and fasting triglycerides | Baseline to 8 days
  These data will be analyzed by fitting mixed effects models for longitudinal data. A model linear in time with random patient intercept and slope effects will be fit initially and residuals examined. If a linear model does not fit the data adequately a quadratic term will be added. Simple paired t-tests of the glucose and triglyceride levels on day 8, 15, and 29 relative to baseline will also be performed.
Change in fasting glucose and fasting triglycerides | Baseline to 15 days
  These data will be analyzed by fitting mixed effects models for longitudinal data. A model linear in time with random patient intercept and slope effects will be fit initially and residuals examined. If a linear model does not fit the data adequately a quadratic term will be added. Simple paired t-tests of the glucose and triglyceride levels on day 8, 15, and 29 relative to baseline will also be performed.
Change in fasting glucose and fasting triglycerides | Baseline to 29 days
  These data will be analyzed by fitting mixed effects models for longitudinal data. A model linear in time with random patient intercept and slope effects will be fit initially and residuals examined. If a linear model does not fit the data adequately a quadratic term will be added. Simple paired t-tests of the glucose and triglyceride levels on day 8, 15, and 29 relative to baseline will also be performed.

SECONDARY OUTCOMES:
Association between genetic variants and changes in fasting glucose and triglycerides | Up to 12 months
  Two-sample t tests will be performed. A Bonferroni adjustment will be applied to control for the number of candidate markers evaluated. Logistic regression models will be fit to determine whether changes in glucose and/or triglycerides are associated with tumor response (complete or partial).
Change in tumor size assessed using RECIST | Up to 2 years
  The change in tumor size will be plotted against the change in glucose/triglyceride and Pearson correlation coefficients will be calculated.
Correlation of toxicities graded using CTCAE version 4.0 with glucose/triglyceride changes | Up to 2 years
  Proportional odds models will be fit to assess whether there is a correlation between toxicities (graded from 0 to 5) and glucose/triglyceride changes.
Regulatory T cells (Tregs) | Baseline to 28 days
  Descriptive statistics will be used to report the quantity and phenotype of Tregs on days 1 and 29 of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Manish R Sharma, MD, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States